CLINICAL TRIAL: NCT02825628
Title: A Randomised, Double-blind, Dose Finding, Repeat Dose Phase II Multicentre Study of ODX for the Treatment of Patients With Castration Resistant Prostate Cancer (CRPC) and Skeletal Metastases
Brief Title: Study of ODX (Osteodex) in Metastatic Castration Resistant Prostate Cancer (CRPC)
Acronym: CRPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DexTech Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ODX-003
Record Dates: First submitted 2016-06-27; First posted 2016-07-07 (Estimated); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer Metastatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Osteodex 3.0 mg/kg (Experimental): formulation: solution for infusion route of administration: intravenous infusion
  Interventions: Drug: Osteodex
- Osteodex 6.0 mg/kg (Experimental): formulation: solution for infusion route of administration: intravenous infusion
  Interventions: Drug: Osteodex
- Osteodex 9.0 mg/kg (Experimental): formulation: solution for infusion route of administration: intravenous infusion
  Interventions: Drug: Osteodex

INTERVENTIONS:
Drug: Osteodex — formulation: solution for infusion route of administration: intravenous infusion
  Other Names: ODX

SUMMARY:
This is a phase II randomised, double-blind, dose finding, repeat dose Phase II multicentre study of ODX for the treatment of patients with castration resistant prostate cancer (CRPC) and skeletal metastases.

The primary objective is to evaluate the relative change from baseline in response markers related to bone metabolism (alkaline phosphatase (B-ALP) and S P1NP) at 12 weeks of three different doses of ODX (3.0, 6.0 and 9.0 mg/kg ODX).

DETAILED DESCRIPTION:
Males, diagnosed with CRPC, who fulfil the inclusion criteria and does not have any exclusion criteria, will be asked to participate in the study. The subject will be informed orally and in writing about the study procedures and give written informed consent, prior to study start.

At the screening visit the following examinations are performed: Physical examination, medical history and concomitant medication. Heart rate, blood pressure, weight, height, body temperature and respiratory rate are measured. Blood samples are drawn and urine sample is collected. ECG is recorded. Bone scan and diagnostic CT scan are also performed. At the next visit, baseline, the subject is examined physically and heart rate, blood pressure, weight, body temperature and respiratory rate are measured, ECG is recorded, blood samples drawn and urine sample collected. FACT-P and EQ-5D-5L (European Quality of Life - 5 Dimensions with 5 levels) questionnaire are filled out by the subject. Adverse events and concomitant medication is documented and the first dose of the investigational product is given.

The subject is surveyed for 3 hours at the hospital.

The duration of the study for the individual subject will be approximately 20 weeks from screening to the follow-up visit 2 weeks after the last dose. Each subject will receive 10 doses of investigational product. After the follow-up visit, the subject enters to long-term follow-up phase which lasts approximately 2 years.

A Data Monitoring Committee (DMC) will be designated and will be responsible to monitor/review all study related safety data. After review of safety data the DMC will provide recommendation as to whether the dose escalation can proceed as planned according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing the informed consent form
2. Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate
3. Evidence of disease progression based on changes in metastatic bone disease (≥2 bone lesions compared to a prior examination) in bone scan and/or other imaging modality AND/OR evidence of PSA progression in the three consecutive determinations at minimum of 1 week intervals
4. Castrate level of serum testosterone ≤1.7 nmol/L
5. Performance status ECOG 0-2
6. Laboratory requirements:

   Haematology:

   Neutrophils ≥ 1.5 x 109/l Haemoglobin ≥ 90 g/l Platelets ≥ 100 x 109/l

   Hepatic function:

   Total S-bilirubin ≤ 1.5 times the upper limit of normal (ULN) AST (SGOT) / ALT (SGPT) ≤ 2.5 times ULN or ≤ 5 times ULN in patients with known liver metastases

   Renal function:

   S-creatinine (S-Cr)≤ 1.5 times ULN
7. No evidence (≤ 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin)
8. Able to adhere to the study visit schedule and other protocol requirements Life expectancy ≥6 months

Exclusion Criteria:

1. Concurrent use of other anti-cancer agents or treatments, with the following exception: a stable dose of Luteinizing Hormone-Releasing Hormone (LHRH) agonist/antagonist or polyestradiol phosphate. Washout period: bicalutamide 6 weeks; flutamide 4 weeks; abiraterone / enzalutamide 6 weeks, chemotherapy 4 weeks; Radium-223 4 weeks; Strontium-89 or Samarium-153 6 months.
2. Any treatment modalities involving palliative radiation therapy or major surgery within 4 weeks prior to treatment in this study
3. Simultaneous participation in any other study involving investigational drugs or having participated in a study less than 4 weeks prior to start of study treatment
4. Any condition, including the presence of laboratory abnormalities, which confounds the ability to interpret data from the study or places the patient at unacceptable risk if he participates in the study
5. Known brain metastases
6. Dental surgery (dental extraction), periodontal disease, local trauma including poorly fitting dentures within 6 months prior to the first dose of study drug
7. Treatment with bisphosphonates or denosumab within 4 weeks prior to first dose of study medication

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-05; Primary Completion 2018-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Relative change from baseline in response markers related to bone metabolism (B-ALP and S P1NP). | Baseline and 20 weeks of treatment

SECONDARY OUTCOMES:
Progression free survival, defined as the time from study entry to the date of disease progression or death from any cause. | Baseline, 20 weeks of treatment and long-term follow-up up to 24 weeks
Overall survival, defined as the time from randomisation to the date of death from any cause. | Baseline, 20 weeks of treatment and long-term follow-up up to 24 weeks
Change from baseline in response markers related to bone metabolism (B-ALP and S P1NP) at each time point sampled (except 12 weeks). | Baseline and 20 weeks of treatment
Change from baseline in response markers related to bone metabolism (Serum C-Terminal Telopeptide (S-CTX) and osteocalcin) at each time point sampled. | Baseline and 20 weeks of treatment
Change from baseline in Prostate Specific Antigen (PSA) at each time point sampled. | Baseline and 20 weeks of treatment
Time to PSA progression | Baseline and 20 weeks of treatment
Time to ALP progression | Baseline and 20 weeks of treatment
Time to P1NP progression | Baseline and 20 weeks of treatment
Time to progression in bone | Baseline and 20 weeks of treatment
Time to progression in soft tissue | Baseline and 20 weeks of treatment
Use of analgesics as reported by the patient during treatment and follow-up | Baseline, 20 weeks of treatment and long-term follow-up up to 24 weeks
Therapy response based on changes from baseline according to Response Evaluation Criteria In Solid Tumors (RECIST) based on diagnostic CT in patients with measurable soft tissue metastases. | Baseline and 20 weeks of treatment
Changes from baseline in bone metastasis by means of bone scan at each time point examined. | Baseline and 20 weeks of treatment
Occurrence of symptomatic skeletal events | Baseline, 20 weeks of treatment and long-term follow-up up to 24 weeks
Pain (FACT-P questionnaire) | Baseline and 20 weeks of treatment
Pain (EQ-5D-5L questionnaire) | Baseline and 20 weeks of treatment
Quality of life (EQ-5D-5L questionnaire) | Baseline and 20 weeks of treatment
Incidence, causality and intensity of Adverse Events (AEs) | Baseline, 20 weeks of treatment and long-term follow-up up to 24 weeks
Dose and duration of medications required for the treatment of AEs | Baseline, 20 weeks of treatment and long-term follow-up up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anders Holmberg, MD, Study Director — DexTech Medical AB
Locations (8):
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Tampere University Hospital, Urology Clinic, Tampere, Finland
- Latvia (2):
  - Latgales Urology Center, Daugavpils
  - Pauls Strandins Clinical University Hospital, Riga
- Sweden (3):
  - Örebro University Hospital, Örebro
  - Urology Clinic, Sodersjukhuset AB, Stockholm
  - Oncology Clinic, Norrlands Universitetssjukhus, Umeå

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thellenberg-Karlsson C, Vjaters E, Kase M, Tammela T, Ojamaa K, Norming U, Nyman C, Andersson SO, Hublarovs O, Marquez-Holmberg M, Castellanos E, Ullen A, Holmberg A, Nilsson S. A randomised, double-blind, dose-finding, phase II multicentre study of ODX in the treatment of patients with castration-resistant prostate cancer and skeletal metastases. Eur J Cancer. 2023 Mar;181:198-207. doi: 10.1016/j.ejca.2022.12.006. Epub 2022 Dec 20. PMID 36682096